CLINICAL TRIAL: NCT05638490
Title: Congenital Talipes Equinovarus Prenatal Diagnosis and Closed Loop Management System Single Center Observational Prospective Study Clinical Study Protocol
Brief Title: Study on Prenatal Diagnosis and Closed-loop Management System of Congenital Talipes Equinovarus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Zhu Xiangyu, Deputy director xiangyu zhu, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: CTE-V1.0
Record Dates: First submitted 2022-11-17; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Prenatal Diagnosis and Closed-loop Management System of Congenital Talipes Equinovarus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — no intervention

SUMMARY:
The study intends to establish a closed-loop management from prenatal to postnatal through prospective cohort, and comprehensively utilize ultrasound and MRI technology to establish a prenatal diagnosis and evaluation system for congenital talipes equinovarus. On the basis of existing genetic testing, further use of whole-exome sequencing and other genomic methods to explore possible pathogenic genes and loci, and clarify the pathogenic mechanism of congenital talipes equinovarus. Therefore, congenital talipes equinovarus can improve its diagnosis and treatment capacity, reduce the disability rate related to congenital talipes equinovarus, and prevent it well.

ELIGIBILITY:
Inclusion Criteria:

1）Single pregnant women 2) "congenital talipes equinovarus" suggested by ultrasound

Exclusion Criteria:

Twin or multiple pregnancies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Single pregnant women with "congenital talipes equinovarus" suggested by ultrasound in our hospital; Voluntary prenatal diagnosis; Those who voluntarily participate in this subject and can comply with the requirements of doctors; Voluntary interview with interviewees:
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Genetic testing results of congenital talipes equinovarus | 2 years
  chromosomal microarray analysis or whole exome screening to find genetic abnormalities of congenital talipes equinovarus

CONTACTS AND LOCATIONS:
Locations (1):
- Drum Tower hospital, Nanjing, Jiangsu, China